CLINICAL TRIAL: NCT06839924
Title: Effect of Motor Cognitive Interference on Cognition and Quality of Life on Multiple Sclerosis Patients
Brief Title: Effect of Motor Cognitive Interference on Cognition and Quality of Life on Patients with Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abd El Aziz, Lecturer Assisstant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T>REC/012/005458
Record Dates: First submitted 2024-12-16; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis, MS
Keywords: Multiple Sclerosis; MS; Cognition; Cognitive Motor Interference; quality of life; Qol
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: external investigator and assessor will be enrolled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Study group will uses Cognitive Motor Interference
  Interventions: Behavioral: Cognitive Motor Interference
- Control group will uses traditional physical therapy (Active Comparator): control group will use traditional physiotherapy
  Interventions: Behavioral: traditional physical therapy

INTERVENTIONS:
Behavioral: Cognitive Motor Interference — Dual task that uses cognitive in addition to Motor training
  Arms: Study group
Behavioral: traditional physical therapy — physiotherapy program including exercises in addition to physical modalities
  Arms: Control group will uses traditional physical therapy

SUMMARY:
Is there an effect of Cognitive Motor Interference on Cognition and quality of life on Multiple Sclerosis patients.

DETAILED DESCRIPTION:
we will assess the effectiveness of Cognitive Motor interference on Cognition and quality of life on Multiple Sclerosis patients

ELIGIBILITY:
Inclusion Criteria:

1. M S patients complain of Mild Cognitive impairment according to Modified Mini Mental State (MMSE).
2. Patients with remission and relapse, primary and secondary progression types of MS.
3. Age between 25 and 45 years.
4. Patients from both gender.

Exclusion Criteria:

1. patients have visual disorders
2. patients have auditory disturbance
3. Non educational patients.
4. Patients with psychiatric disorders.
5. Patients with mod to severe cognitive impairment according to MMSE

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Cognition (working memory and divided attention) | baseline assessment and after 12 sessions of Cognitive motor interference 3 sessions per weak for 4 weaks
  cognition domains including working memory and divided attention will be assessed by rehacom V 6.10.2.0 software

SECONDARY OUTCOMES:
A health-related quality of life | Baseline assessment and after 12 sessions of Cognitive motor interference 3 sessions per weak for 4 weaks
  quality of life will be assessed by Multiple Sclerosis Quality of Life (MSQOL)-54 Instrument

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No